CLINICAL TRIAL: NCT04852445
Title: The Temporal Cellular Landscape of the Adaptive Immune System in Patients With Acute Stroke
Acronym: TAPAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Diederik van de Beek, The temporal cellular landscape of the adaptive immune system in patients with acute stroke, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: TAPAS
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, lymphoid tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stroke: We will include: 60 patients aged 18 years or older with clinical symptoms of hemispheric ischemic stroke due to occlusion of a large cerebral blood vessel, onset within 48 hours and NIHSS of 1 or more;
- Controls: 30 healthy controls, age- and sex- matched with stroke study population
- Carotid arterectomy after stroke: 10 patients undergoing carotid endarterectomy within 30 days after stroke
- Carotid endarterectomy for asymptomatic stenosis: 3 patients without stroke undergoing carotid endarterectomy for asymptomatic carotid stenosis.

SUMMARY:
Despite novel acute therapies the global burden of stroke remains high worldwide. Targeting the immune response after stroke has the potential to improve recovery in all stroke patients. Experimental studies suggest important roles for T-lymphocytes, especially anti-inflammatory regulatory T cells, in the evolution of stroke and neurological deficit. Objectives of this study are to either confirm or refute the hypothesis that a subset of brain regulatory T cells exists in humans and expands after stroke and to identify immunological biomarkers that can be used in stroke clinical trials targeting the adaptive immune system.

DETAILED DESCRIPTION:
Rationale: despite novel acute therapies the global burden of stroke remains high worldwide. Targeting the immune response after stroke has the potential to improve recovery in all stroke patients. Experimental studies suggest important roles for T-lymphocytes, especially anti-inflammatory regulatory T cells, in the evolution of stroke and neurological deficit.

Objective:

1. To confirm that patients experience an increase and migration of CD4+CD25+FoxP3+ "brain" Tregs..
2. To characterize and subgroup brain T reg cells; to assess clonality of the T reg cells in order to determine whether a specific antigen-reaction is present; to assess whether specific antigen-directed FoxP3+ brain Treg cells are recruited through cervical lymph nodes and subsequently migrate towards the brain; to assess whether T reg cells play a role in neurotoxic astrogliosis after stroke.

Study design: case control study.

Study population: we will include: 60 patients aged 18 years or older with clinical symptoms of hemispheric ischemic stroke due to occlusion of a large cerebral blood vessel, onset within 48 hours and NIHSS of 1 or more; 30 healthy age- and sex- matched controls; 10 patients undergoing carotid endarterectomy within 30 days after stroke and 3 patients without stroke undergoing carotid endarterectomy for asymptomatic carotid stenosis.

Main study parameters/endpoints: we will assess the amount and characteristics of regulatory T cells in peripheral blood and lymph nodes and compare these with patients without stroke.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: in 60 patients blood will be sampled at 9 time points. In addition, neurologic examination at 5 time points, 1 MRI scan and 1 telephone interview will be performed. In 10 patients who undergo carotid endarterectomy, a lymph node will be extracted and blood will be drawn during this surgery. The study is carried out in both capacitated and incapacitated persons because exclusion of non-communicative stroke patients would lead to a selective patient sample.

ELIGIBILITY:
Inclusioncriteria

In order to be eligible to participate in part 1 of this study (serial blood sampling), a subject must meet all of the following criteria:

* age 18 years or older,
* clinical symptoms of hemispheric ischemic stroke due to occlusion of a large vessel
* an onset of symptoms less than 48 h
* a score of 1 or more on the National Institutes of Health Stroke Scale (NIHSS)
* admission to hospital
* written informed consent obtained

For the control arm of part 1 of the study:

* age 18 years or older
* increased risk of cardiovascular disease (defined as a previous cardiovascular event other than stroke or one of the following risk factors: smoking, hypertension, hypercholesterolemia or diabetes mellitus)
* written informed consent obtained
* scheduled blood draw ordered at the Neurology outpatient clinic at Amsterdam UMC (location AMC) for non-vascular non-immunological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: we will include: 60 patients aged 18 years or older with clinical symptoms of hemispheric ischemic stroke due to occlusion of a large cerebral blood vessel, onset within 48 hours and NIHSS of 1 or more; 30 healthy age- and sex- matched controls; 10 patients undergoing carotid endarterectomy within 30 days after stroke and 3 patients without stroke undergoing carotid endarterectomy for asymptomatic carotid stenosis.
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Regulatory T cells | 28 days
  we will assess the amount and characteristics of regulatory T cells in peripheral blood and lymph nodes and compare these with patients without stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic University Medical Center Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided